CLINICAL TRIAL: NCT02427321
Title: Cystoscopic Imaging Collection and Enhancement pROject: A Prospective, Non-randomised, Observational Proof-of-concept Study of Flexible Cystoscopic Examination Recordings From a Symptomatic Adult Population
Brief Title: Cystoscopic Imaging Collection and Enhancement pROject
Acronym: CICERO
Status: Completed | Type: Observational
Sponsor: Biosignatures Limited (Industry)
Collaborators: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: PR-14056
Record Dates: First submitted 2015-04-17; First posted 2015-04-28 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Urinary Bladder Neoplasms
Keywords: Cystoscopy; Bladder cancer; Bladder imaging
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cystoscopy cohort: Video recording of flexible cystoscopic examination. All participants enrolled on the study will have video from their flexible cystoscopic examination recorded.
  Diagnosis and pathology information will be collected from the participants medical notes for a period of eight weeks following the recorded cystoscopy.
  Interventions: Device: Video recording of flexible cystoscopic examination

INTERVENTIONS:
Device: Video recording of flexible cystoscopic examination — The video feed from the flexible cystoscopic examination will be recorded for all participants in the study. Proof-of-concept device will record high-definition video in a lossless format to a computer hard-drive from any existing cystoscopy equipment

SUMMARY:
This study will collect video recordings of routine flexible cystoscopy examinations, medical history and diagnosis information, from up to 100 participants who have a history of bladder cancer, or symptoms suggestive of bladder cancer, in order to develop a new computer system for recording and reviewing images of the bladder, and to assess the utility of this system.

DETAILED DESCRIPTION:
Flexible cystoscopy is commonly used in the diagnosis and post-treatment care of bladder cancer, the 7th most common cancer in the United Kingdom. While the equipment to record bladder examinations exists, it is not simple or quick to use so examinations are rarely recorded. Methods of enhancing the images obtained during these examinations also exist but these are generally hardware based, requiring specific equipment, or use a fluorescent dye and special endoscope, which is expensive for the clinical service provider, inconvenient for the patient and may cause allergic reactions.

The new proof-of-concept device will record high-definition video in a lossless format to a computer hard-drive from any existing cystoscopy equipment to which it can be connected. Additionally, the device incorporates a foot pedal which allows the operator to "bookmark" points of interest during the examination. These points are marked in the recorded video data file and aid later navigation and review of examination session videos.

The recordings will be used to develop novel image enhancement software, which is intended to make abnormalities in the bladder easier to identify. Once the software has been developed, the enhanced and un-enhanced videos will be reviewed by experts (clinical urology specialists) and non-experts (other healthcare staff and laypeople), who will be asked to report areas of interest in the videos, without knowledge of the diagnosis for each examination. A statistical analysis of reporting of areas of interest by expert and non-expert reviewers will be produced, to assess the usefulness of the software image enhancement in identifying abnormalities in the bladder.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled to undergo cystoscopy examination as they are considered to possibly have undiagnosed bladder cancer, or;
* patients scheduled to undergo a post-treatment follow-up or routine surveillance cystoscopy examination, having previously been treated for bladder cancer; and
* Have provided written informed consent agreeing to participation in the study prior to any study-specific procedures being carried out.

Exclusion Criteria:

* patients who are incapable of providing written informed consent agreeing to participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults referred to Urology clinic for cystoscopic surveillance after treatment for bladder cancer, and adults referred for cystoscopic investigation of haematuria or lower urinary tract symptoms (LUTS) that raise the suspicion of an undiagnosed bladder cancer.
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2015-05; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Video recording of cystoscopic examination and diagnosis | As time of cystoscopic examination - Visit 1, day 1, diagnostic and pathology information collected for up to 8 weeks following Visit 1
  A set of high quality recorded cystoscopy examinations from 50 to 100 participants. The recordings will be used to develop novel image enhancement software, which is intended to make abnormalities in the bladder easier to identify. The diagnosis reported by the cystoscope operator will be reported at the time of the examination. Pathology derived diagnosis and any other additional information regarding the diagnosis and subsequent treatment will be recorded at 8 weeks following the initial examination (Visit 1, day 1).

SECONDARY OUTCOMES:
Expert opinions of clinical team | Reported following recording of all cystoscopic examinations - approximately 3 months following recruitment of first participant
  Written expert opinions from the clinical team based on structured review of a subset of the recordings in raw and enhanced playback modes, including comments on the quality of the recordings made by the device and their suitability for use as a documentary record of the examination procedure.
Statistical summary | Once data collection from all participants is complete - approximately 5 months after first patient is recruited
  A statistical summary of the inter-observer consistency in reporting 'areas of interest' in raw and enhanced video sequences. This will report on expert and non-expert reviewer results.
Report on 2 and 3 (correspondence between the results of 2) expert opinion and 3)statistical summary, and the diagnostic outcomes logged by the clinic. | Once data collection is complete - approximately 5 months after first patient is recruited
  A report exploring the correspondence between the results of 2) and 3) and the diagnostic outcomes logged by the clinic.
Expert opinion on usability and reliability | Once data collection is complete - approximately 5 months after first patient is recruited
  Written expert opinions from the clinical team which will comment on the usability and reliability of the device compared to existing recording and documenting systems, including whether use of the device has any adverse impact upon patient safety caused by an increase in the duration or disruption of routine cystoscopy procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh Heer, PhD FRCS, Principal Investigator — Newcastle University, NICR